CLINICAL TRIAL: NCT05801276
Title: Exploration of Plasma CDO1 and HOXA9 DNA Methylation for Detecting Epithelial Ovarian Cancer: A Clinical Trial in China
Brief Title: ctDNA Methylation for Detecting Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-METHY2
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Epithelial Ovarian Cancer; Circulating Tumor DNA; DNA Methylation; Non-invasive Diagnosis; CA125; Human Epididymis Protein 4; ROMA Index; Imaging Evaluation; Survival Prognosis
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma circulating tumor DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Methylation assay — Methylation assay of CDO1 and HOXA9 genes in plasma circulating tumor DNA

SUMMARY:
Ovarian cancer is one of the most dangerous and leading gynecological cancer, with significant cancer-related mortality among women. However, current detection methods are still limited, with approximately 70% of patients with high-grade serous ovarian cancer often being advanced at the initial diagnosis and more than 80% with intraperitoneal spread. The five-year survival rate for late detection is only 29%; on the contrary, if detected early, the five-year survival rate can reach 92%. Therefore, early diagnosis and detection are essential in diagnosing and treating ovarian cancer. Liquid biopsy has attracted widespread attention because of its non-invasive, real-time, and dynamic characteristics. Cell-free DNA in plasma can identify a small tumor burden well and reflect the clinical cancer information of cells.The role of hypermethylation in developing malignant tumors has received increasing attention. Methylation is one of epigenetics and plays a vital role in the occurrence and development of tumors. According to previous research basis of the researchers, it has been found that CDO1 and HOXA9 genes show hypermethylation in ovarian cancer, and they are considered one of the biomarkers for detection. Therefore, this study will further explore the detection of CDO1 and HOXA9 methylation levels based on cell-free DNA in blood and compared with ovarian pathology results; the application of methylation detection technology in ovarian cancer/precancerous lesions will further explore the application value of non-invasive diagnosis and prognostic follow-up.This study will involve three centers and is expected to enroll more than 1,400 clinical subjects, further examine the consistency of methylation detection kits with the histopathological examination, ROMA index, and Sanger sequencing results, and obtain sensitivity and specificity technical performance parameters.

DETAILED DESCRIPTION:
This study has two phases: the "Clinical Performance Validation" cohort and the "Assay Accuracy Verification" cohort.

The " Clinical Performance Validation" phase of this study will assess the reagents to detect plasma samples; patients undergo routine examinations by clinical trial institutions, including but not limited to tumor markers and histopathological examinations. The clinical performance of the assessment reagents was systematically evaluated by evaluating the consistency between the test results of the assessment reagents and the histopathological examination results, as well as the surface of the ROMA index and the histopathological examination results.

During the "Assay Accuracy Verification" phase of this study, a part of the qualified samples was randomly selected. The Sanger sequencing method was used as a comparison method to evaluate the detection accuracy of the test reagents for detecting the methylation of CDO1 and HOXA9 genes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ready for surgical treatment for pelvic mass or adnexal mass
* Age is greater than or equal to 18 years
* Not receiving any chemotherapy, physical therapy, or surgical treatment for ovarian lesions
* With ovarian pathology
* Willing to be tested and signed an informed consent form
* With available data of plasma CA125, Human epididymis protein 4 and effective imaging results
* The study will also enroll several patients with primary breast cancer, lung cancer, colon cancer, uterine cervical cancer and uterine carcinomas

Exclusion Criteria:

* Not meeting all the including criteria
* A sample of patients withdrawing from the trial
* Samples that the investigator believes should be excluded from this trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ready for surgical treatment for pelvic mass or adnexal mass. The study will also enroll several patients with primary breast cancer, lung cancer, colon cancer, uterine cervical cancer and uterine carcinomas.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity | One month
  Diagnostic sensitivity of methylation assay for detecting epithelial ovarian cancer
Diagnostic specificity | One month
  Diagnostic specificity of methylation assay for detecting epithelial ovarian cancer

SECONDARY OUTCOMES:
Progression-free survival | Two years
  Progression-free survival after the last treatment for cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China